CLINICAL TRIAL: NCT01145456
Title: A Phase I Study of R04929097 in Combination With Gemcitabine in Patients With Advanced Solid Tumors
Brief Title: Gamma-Secretase Inhibitor RO4929097 and Gemcitabine Hydrochloride in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01433; NCI-2011-01433 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000674950; PHL-078 (Other: University Health Network-Princess Margaret Hospital); 8575 (Other: CTEP); U01CA132123 (NIH); NCT01189539 (obsolete NCT alias)
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2013-12

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; Gemcitabine

ARMS (1):
- Treatment (RO4929097 and gemcitabine hydrochloride) (Experimental): Patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-3, 8-10, 15-17, and 22-24 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Drug: gemcitabine hydrochloride; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097 — Given orally
  Other Names: R4733; RO4929097
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of gamma-secretase inhibitor RO4929097 when given together with gemcitabine hydrochloride in treating patients with advanced solid tumors. Gamma-secretase inhibitor RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving gamma-secretase inhibitor RO4929097 together with gemcitabine hydrochloride may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety profile and establish the maximum-tolerated dose and recommended phase II dose of gamma-secretase inhibitor RO4929097 in combination with gemcitabine hydrochloride in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetic profile of gamma-secretase inhibitor RO4929097 when given in combination with gemcitabine hydrochloride and to correlate the pharmacokinetic profile with toxicity and biological activity.

II. To assess the antitumor activity of gamma-secretase inhibitor RO4929097 and gemcitabine hydrochloride in patients with advanced solid tumors.

III. To correlate the expression of biomarkers of Notch signaling in archival tumor tissue with antitumor activity of gamma-secretase inhibitor RO4929097 in combination with gemcitabine hydrochloride.

OUTLINE: This is a multicenter, dose-escalation study of gamma-secretase inhibitor RO4929097.

Patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-3, 8-10, 15-17, and 22-24 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Plasma and blood samples may be collected periodically for pharmacokinetic studies and biomarker analysis.

After completion of study treatment, patients are followed up every 1 month for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Meets one of the following sets of criteria:

  * Histologically and/or cytologically confirmed solid malignancy

    * Metastatic or unresectable disease
    * Disease for which standard curative or palliative measures do not exist or are no longer effective
  * Histologically and/or cytologically confirmed adenocarcinoma of the pancreas (for patients in the expansion cohort)

    * Locally advanced or metastatic disease
    * No prior chemotherapy for advanced disease
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan
* No known brain metastases
* ECOG performance status (PS) 0-1 (Karnofsky PS 60-100%)
* Life expectancy > 12 weeks
* Hemoglobin ≥ 90 g/L (or ≥ 9 g/dL)
* Leukocytes ≥ 3,000/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 1.25 times upper limit of normal (ULN)
* AST/ALT ≤ 1.5 times ULN
* Serum creatinine =< ULN OR creatinine clearance ≥ 60 mL/min
* No uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia, or hypokalemia, defined as less than the lower limit of normal despite adequate electrolyte supplementation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use two forms of adequate contraception (i.e., barrier contraception and one other method of contraception) for ≥ 4 weeks before, during, and for ≥ 12 months after completion of study treatment
* Able to swallow medication
* No malabsorption syndrome or other condition that would interfere with intestinal absorption
* No uncontrolled concurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia other than chronic, stable atrial fibrillation
  * Psychiatric illness or social situations that would limit compliance with study requirements
* No baseline QTc > 450 msec (for male patients) or > 470 msec (for female patients)
* No history of risk factors for QT interval prolongation including, but not limited to, a family or personal history of any of the following:

  * Long QT syndrome
  * Recurrent syncope without known etiology
  * Sudden unexpected death
* No history of torsade de pointes or other significant cardiac arrhythmias or the need for concomitant meds with known potential to prolong QT interval or antiarrhythmics
* No diarrhea ≥ grade 2 not under control with standard anti-diarrhea medications
* No serologic positivity for hepatitis A, B, or C
* No history of liver disease or other forms of hepatitis or cirrhosis
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to gamma-secretase inhibitor RO4929097 or to gemcitabine hydrochloride
* Female patients may not donate ova during or after completion of study treatment
* Male patients may not donate sperm during and for ≥ 12 months after completion of study treatment
* Patients may not donate blood during and for ≥ 12 months after completion of study treatment
* No other concurrent investigational or commercial agents or therapies administered with the intent to treat the patient's malignancy
* Any number of prior therapies allowed
* No prior therapy with a Notch inhibitor
* At least 4 weeks since prior radiotherapy, chemotherapy, or systemic therapy (6 weeks if the last regimen included nitrosourea or mitomycin C) and recovered

  * Exceptions may be made for low-dose, non-myelosuppressive radiotherapy for symptomatic palliation
* Patients in the expansion cohort must meet the following criteria:

  * No prior chemotherapy for advanced disease except for fluorouracil (with or without folinic acid) or gemcitabine hydrochloride given concurrently with radiotherapy as a "radiosensitizer"
  * At least 6 months since prior adjuvant gemcitabine hydrochloride
  * Prior radiotherapy for the management of local disease allowed provided > 4 weeks have elapsed since the last radiation treatment and all toxicities have resolved
  * Patients who have had radiotherapy to their sole site of disease are eligible provided they have documented progression of that lesion before study registration
* Recovered from side effects of previous systemic anticancer therapy to ≤ CTCAE grade 2
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®)
* No concurrent medications with known potential to prolong QT interval
* No concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4
* No concurrent medications or food that may interfere with the metabolism of gamma-secretase inhibitor RO4929097, including ketoconazole and grapefruit or grapefruit juice
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-06; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of RO4929097 in combination with gemcitabine hydrochloride, defined as the dose level in which no more than 1 of 6 patients or 0/3 experience DLT, graded according to NCI CTCAE version 4.0 | 28 days

SECONDARY OUTCOMES:
Cmax, Tmax, t 1/2, AUC0-24, and clearance of gamma-secretase/Notch signalling pathway inhibitor RO4929097 and gemcitabine hydrochloride when given together | Before dosing and at 1, 2, 4, 6, 8, and 24 hours after dosing on days 1 and 10; before dosing on days 3, 9, and 15; before dosing and 1 and 2 hours after dosing on day 8; and any time on day 22 of course 1 and before drug dosing on day 1 of course 2
Objective response according to RECIST criteria 1.1 | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bedard, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (2):
- Canada (2):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario